CLINICAL TRIAL: NCT02984319
Title: Effect of Cherry Concentrate on Vascular Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Exeter (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 115229/03
Record Dates: First submitted 2016-12-02; First posted 2016-12-06 (Estimated); Last update posted 2018-10-25 (Actual); Status verified 2018-10

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cherry (Active Comparator): Cherry concentrate
  Interventions: Dietary Supplement: Cherry versus placebo concentrate
- Placebo (Placebo Comparator): Placebo concentrate
  Interventions: Dietary Supplement: Cherry versus placebo concentrate

INTERVENTIONS:
Dietary Supplement: Cherry versus placebo concentrate — Acute cherry concentrate

SUMMARY:
Acute effect of cherry concentrate consumption on flow mediated dilatation in healthy young men

ELIGIBILITY:
Inclusion Criteria:

* no prescription medications

Exclusion Criteria:

* prescription medications

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2015-11; Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Flow mediated dilatation | Change from baseline to 3 hours post dietary supplementation

SECONDARY OUTCOMES:
Microvascular function (laser doppler flowmetry) | Change from baseline to 3 hours post dietary supplementation
Plasma nitrite concentration | Change from baseline to 3 hours post dietary supplementation

CONTACTS AND LOCATIONS:
Locations (1):
- Sport & Health Sciences, Exeter, Devon, United Kingdom

IPD SHARING:
Plan to Share IPD: No